CLINICAL TRIAL: NCT06812780
Title: A Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD2389 (CAMPOLINA)
Brief Title: A Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of AZD2389
Acronym: CAMPOLINA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D7930C00004
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Impairment
Keywords: Mild; Moderate; Severe; Matched Healthy Controls; Liver Fibrosis; Liver Cirrhosis
MeSH Terms: conditions — Lymphoma, Follicular; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled within the following groups based on their CP classification score as determined at screening: Cohort 1: Participants with normal hepatic function (sex-, age-, and body mass index [BMI]-matched)
  * Cohort 2: Participants with mild hepatic impairment (CP A classification)
  * Cohort 3: Participants with moderate hepatic impairment (CP B classification)
  * Cohort 4 (Optional): Participants with severe hepatic impairment (CP C classification)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants with normal hepatic function (sex-, age-, and body mass index [BMI]-matched)
  Interventions: Drug: AZD2389
- Cohort 2 (Experimental): Participants with mild hepatic impairment (CP A classification)
  Interventions: Drug: AZD2389
- Cohort 3 (Experimental): Participants with moderate hepatic impairment (CP B classification)
  Interventions: Drug: AZD2389
- Cohort 4 (Experimental): Participants with severe hepatic impairment (CP C classification)
  Interventions: Drug: AZD2389

INTERVENTIONS:
Drug: AZD2389 — Single oral dose of AZD2389 in participants from all cohorts

SUMMARY:
The purpose of this study is to examine the safety and tolerability of AZD2389 in participants with hepatic impairment and participants with normal hepatic function.

DETAILED DESCRIPTION:
This is a single-dose, non-randomised, open-label, parallel-group study to examine the PK, fibroblast activation protein activity, safety, and tolerability of AZD2389 in participants with hepatic impairment and participants with normal hepatic function.

The study is planned to consist of:

* Cohort 1: Participants with normal hepatic function (sex-, age-, and body mass index [BMI]-matched)
* Cohort 2: Participants with mild hepatic impairment (CP A classification)
* Cohort 3: Participants with moderate hepatic impairment (CP B classification)
* Cohort 4 (Optional): Participants with severe hepatic impairment (CP C classification)

Safety, tolerability, and available plasma PK data up to 48 hours post-dose from at least 4 participants in each of the mild hepatic impairment (CP Class A) and moderate hepatic impairment (CP Class B) cohorts must have been assessed by the investigator(s), medical monitor, and sponsor prior to the decision to proceed with evaluation/recruitment of participants with severe hepatic impairment (CP Class C). Cohort 1 (normal hepatic function) will be initiated in parallel with Cohorts 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

For Hepatic:

* Participant with a diagnosis of stable hepatic impairment

For Healthy:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.

All participants:

- Body weight ≥ 50 kg; BMI within the range of 18.0 to 42.0 kg/m2 (inclusive).

Exclusion Criteria:

* Participant has eGFR < 60 mL/minute/1.73 m2
* Positive test for HIV at screening
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity
* History of severe dermatological disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Plasma PK parameter Cmax | pre-dose to 48 hours post-dose
  maximum observed plasma concentration
Plasma PK parameter AUCinf | pre-dose to 48 hours post-dose
  area under the concentration-time curve from zero to infinity
Plasma PK parameter AUClast | pre-dose to 48 hours post-dose
  area under the concentration-time curve from zero to the last measurable concentration

SECONDARY OUTCOMES:
Plasma PK parameter t1/2λz | pre-dose to 48 hours post-dose
  half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve
Plasma PK parameter Tmax | pre-dose to 48 hours post-dose
  time to reach maximum observed plasma concentration
Plasma PK parameter CL/F | pre-dose to 48 hours post-dose
  apparent total body clearance of drug from plasma after extravascular administration
Plasma PK parameter Vz/F | pre-dose to 48 hours post-dose
  apparent volume of distribution during the terminal phase after extravascular administration.
Urine PK parameter Ae(t1-t2) | pre-dose to 48 hours post-dose
  cumulative amount of unchanged drug excreted into the urine for the interval between time 1 and time 2
Urine PK parameter CLr | pre-dose to 48 hours post-dose
  renal clearance of the drug from plasma
Urine PK parameters fe(t1-t2) | pre-dose to 48 hours post-dose
  fraction of the drug excreted into the urine for the interval between time 1 and time 2

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Chandler, Arizona
  - Research Site, Rialto, California
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida
  - Research Site, San Antonio, Texas